CLINICAL TRIAL: NCT02771795
Title: A Long-term Follow-up Study for Cardiac Safety in the Patients With HER2 Positive Early or Locally Advanced Breast Cancer Who Have Completed the SB3-G31-BC
Brief Title: A Long-term Follow-up Study for Cardiac Safety in the Patients With HER2 (+) Breast Cancer Who Have Completed the SB3-G31-BC
Status: Terminated | Type: Observational
Why Stopped: Considering the life-threatening risk posed by COVID-19 disease to a fragile population, the Sponsor concluded that the benefit of continuing the study does not outweigh the risk to the safety of patients & site staffs.
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SB3-G31-BC-E
Record Dates: First submitted 2016-05-09; First posted 2016-05-13 (Estimated); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Breast Neoplasms
Keywords: HER2; Trastuzumab; Biosimilar; Cancer; Breast; Positive
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Herceptin (trastuzumab): Intravenous administration
  Interventions: Drug: Herceptin (trastuzumab)
- SB3 (proposed trastuzumab biosimilar): Intravenous administration
  Interventions: Drug: SB3 (proposed trastuzumab biosimilar)

INTERVENTIONS:
Drug: Herceptin (trastuzumab) — Intravenous administration
  Other Names: Herceptin
  Groups: Herceptin (trastuzumab)
Drug: SB3 (proposed trastuzumab biosimilar) — Intravenous administration
  Groups: SB3 (proposed trastuzumab biosimilar)

SUMMARY:
A Long-term Follow-up Study for Cardiac Safety in the Patients with HER2 Positive Early or Locally Advanced Breast Cancer Who Have Completed the SB3-G31-BC

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received the study treatment of SB3-G31-BC.
* Subjects who provide informed consent.

Exclusion Criteria:

* Subjects unwilling to follow the study requirements are not eligible for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2 positive early or locally advanced breast cancer who received SB3 or Herceptin according to clinical trial SB3-G31-BC.
Sampling Method: Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2016-04; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- Complex Oncological Center - Vratsa, EOOD, Vratsa, Bulgaria
- ONKOCENTRUM Medicon Services s.r.o., Prague, Czechia
- France (2):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Centre Hospitalier de Belfort-Montbeliard, Montbéliard
- Poland (8):
  - Bialostockie Centrum Onkologii im.M.Sklodowskiej-Curie w Bialymstoku, Bialystok
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii I Radioterapii, Gdansk
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej, Olsztyn
  - Samodzielny Publiczny ZOZ Opolskiego Centrum Onkologii w Opolu im. T. Koszarowskiego, Opole
  - Wielkopolskie Centrum Onkologii, im Marii Sklodowskiej-Curie, Poznan
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw
  - Magodent Sp. Z o.o., Warsaw
- Romania (8):
  - Spitalul Judetean de Urgenta "Dr. Constantin Opris" Baia Mare, Baia Mare
  - SC Centrul Medical Unirea SRL-Policlinica Baneasa, Specialitatea Oncologie Medicala, Bucharest
  - Spitalul Clinic Filantropia, Compartimentul Oncologie Ginecologica, Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
  - Spitalul Municipal Ploiesti, Sectia Oncologie Medicala, Ploieşti
  - S.C Oncomed S.R.L, Timișoara
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Russia (11):
  - SBHI of Moscow City "Moscow City Oncology Hospital №62" of Moscow Healthcare Department, Istra, Krasnogorsk District
  - S.I. Russian Oncological Research Center n.a. N.N. Blokhin, Moscow
  - Federal State Budgetary Institution "Federal Medical Research Center n.a. P.A Gertsen" of Ministry of healthcare of RF/3, Moscow
  - SBI of Ryazan region "Regional Clinical Oncological Dispensary", Ryazan
  - SBHI "Leningrad Regional Oncology Dispensary", Saint Petersburg
  - Non-state Healthcare Institution "Roadway Clinical Hospital of OJSC Russian Railways", Saint Petersburg
  - Saint-Petersburg SBHI "City Clinical Oncology Dispensary", Saint Petersburg
  - FSI "Scientific and Research Institution of Oncology n.a. N.N.Petrov" of Ministry of Healthcare and SD of RF, Saint Petersburg
  - SBHI "Saint-Petersburg Scientific and Practical Center of Specialized Methods of Medical Help (oncological), Saint Petersburg
  - SHBI of Yaroslavl Region "Regional Clinical Oncology Hospital", Yaroslavl
  - BHI of Omsk Region "Clinical Oncology Dispensary", Оmsk
- Ukraine (9):
  - Communal Institution Cherkasy Regional Oncological Dispensary of Cherkasy Regional Council, Cherkasy
  - Communal Institution Dnipropetrovsk City Multifield Clinical Hospital No.4 of Dnipropetrovsk Regional Council, Dnipropetrovsk
  - Communal Non-commercial Enterprise Regional Center of Oncology, Kharkiv
  - Communal Institution of Kherson Regional Council Kherson Regional Oncological Dispensary, Kherson
  - Lviv State Oncological Regional Treatment and Diagnostic Center, Lviv
  - Regional Communal Institution Sumy Regional Clinical Oncological Dispensary, Sumy
  - Uzhgorod Central City Clinical Hospital City Oncological Center, Uzhhorod
  - Vinnytsia Regional Clinical Oncological Dispensary, Vinnytsia
  - Communal Institution Zaporizhzhia Regional Clinical Oncological Dispensary of Zaporizhzhia Regional Council, Zaporizhzhia

REFERENCES:
- [Derived] Pivot X, Cortes J, Luftner D, Lyman GH, Curigliano G, Bondarenko IM, Ahn JH, Im SA, Litwiniuk M, Shparyk YV, Ho GF, Kislov NV, Wojtukiewicz M, Sarosiek T, Chae YS, Ahn JS, Jang H, Kim S, Lee J, Yoon Y. Cardiac Safety and Efficacy of SB3 Trastuzumab Biosimilar for ERBB2-Positive Early Breast Cancer: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e235822. doi: 10.1001/jamanetworkopen.2023.5822. PMID 37022687
- [Derived] Pivot X, Pegram M, Cortes J, Luftner D, Lyman GH, Curigliano G, Bondarenko I, Yoon YC, Kim Y, Kim C. Three-year follow-up from a phase 3 study of SB3 (a trastuzumab biosimilar) versus reference trastuzumab in the neoadjuvant setting for human epidermal growth factor receptor 2-positive breast cancer. Eur J Cancer. 2019 Oct;120:1-9. doi: 10.1016/j.ejca.2019.07.015. Epub 2019 Aug 21. PMID 31445454

RESULTS

PARTICIPANT FLOW:
Groups:
- Herceptin (Trastuzumab): Intravenous administration
  Herceptin (trastuzumab): Intravenous administration in SB3-G31-BC study (NCT02149524). No additional IP was administered for this study since it was an observational study.
- SB3 (Proposed Trastuzumab Biosimilar): Intravenous administration
  SB3 (proposed trastuzumab biosimilar): Intravenous administration in SB3-G31-BC study (NCT02149524). No additional IP was administered for this study since it was an observational study.
Period: Overall Study
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar)
Started | 271 | 267
Completed | 56 | 45
Not Completed | 215 | 222
Not completed — Withdrawal by Subject | 47 | 37
Not completed — Termination by premature discontinuation of study | 168 | 185

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar) | Total
Number analyzed (Participants) | 271 | 267 | 538
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 266 | 262 | 528
  >=65 years | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 271 | 267 | 538
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 270 | 266 | 536
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Asymptomatic Significant LVEF Decrease
Description: Asymptomatic significant LVEF decrease is defined as LVEF decline ≥ 10% points from baseline and resulting LVEF < 50%
Time Frame: approximately 56 months (median follow-up duration)
Population: Long-term follow-up set
Measure: Count of Participants; unit: Participants
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar)
Number analyzed (Participants) | 181 | 186
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Through end of the study, approximately 4.7 years; Since SB3-G31-BC-E study was to assess the long-term cardiac safety for SB3 or Herceptin®, which was mainly about post-dose cardiac toxicities captured through cardiac assessments, non-serious AEs were not intended to be collected through this study.
Description: For any type of serious AE (SAE; cardiac or non-cardiac) that could be determined by the Investigator to be related to the IP then that SAE was reported through a separate paper SAE report form to the Sponsor.
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar)
All-Cause Mortality (participants affected / at risk) | 38/271 | 22/267
Serious Adverse Events (participants affected / at risk) | 1/271 | 0/267
Other Adverse Events (participants affected / at risk) | 0/271 | 0/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Herceptin (Trastuzumab) (N=271) | SB3 (Proposed Trastuzumab Biosimilar) (N=267)
cardiac death (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
- At least sixty (60) dayas prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy of all such manuscripts and materials, and allow the Sponsor sixty (60) days to review and comment on them to ensure that the publication would not disclose any Confidential Information or impair the Sponsor's ability to obtain patent protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT02771795/Prot_SAP_000.pdf